CLINICAL TRIAL: NCT05369403
Title: An Open-Label, Study to Evaluate the Safety and Efficacy of Lebrikizumab in Adult and Adolescent Participants With Moderate-to-Severe Atopic Dermatitis Previously Treated With Dupilumab
Brief Title: A Study of Lebrikizumab (LY3650150) in Adult and Adolescent Participants With Moderate-to-Severe Atopic Dermatitis Previously Treated With Dupilumab
Acronym: ADapt
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18499; J2T-MC-KGBO (Other: Eli Lilly and Company)
Record Dates: First submitted 2022-05-06; First posted 2022-05-11 (Actual); Results first posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Atopic Dermatitis
Keywords: Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — lebrikizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lebrikizumab (Experimental): Participants will receive Lebrikizumab by subcutaneous (SC) injection.
  Interventions: Drug: Lebrikizumab

INTERVENTIONS:
Drug: Lebrikizumab — Administered SC
  Other Names: LY3650150; DRM06

SUMMARY:
The study will assess the safety and efficacy of lebrikizumab in adult and adolescent participants with moderate-to-severe atopic dermatitis (AD) previously treated with Dupilumab.

ELIGIBILITY:
Inclusion Criteria:

* All participants must have prior treatment with dupilumab meeting one of the following conditions:

  * Participants who stopped dupilumab treatment due to non-response, partial response, loss of efficacy must have been previously treated with dupilumab (at labeled dose level) for at least 4 months.
  * Participants who stopped dupilumab treatment due to intolerance or adverse events (AEs) to the drug may enter the study with no required prior length of dupilumab treatment.
  * Participants who stopped dupilumab treatment due to cost or loss of access to dupilumab (for example, insurance coverage) may enter the study with no required prior length of dupilumab treatment.
* Participants who have chronic AD that has been present for ≥1 year before screening.
* Have EASI ≥16 at baseline
* Have IGA score ≥3 (Scale of 0 to 4) at baseline
* Have ≥10% body surface area (BSA) of AD involvement at baseline
* Have a history of inadequate response to treatment with topical medications; or determination that topical treatments are otherwise medically inadvisable.
* Adolescents body weight must be ≥40 kg at baseline.

Exclusion Criteria:

* History of human immunodeficiency virus (HIV) infection or positive HIV serology at screening.
* Have a current infection or chronic infection with hepatitis B virus (HBV) at screening (that is, positive for hepatitis B surface antigen and/or polymerase chain reaction positive for HBV DNA
* Have a current infection with hepatitis C virus (HCV) at screening (that is, positive for HCV RNA
* Have an uncontrolled chronic disease that might require multiple intermittent uses of oral corticosteroids at screening, as defined by the investigator.
* Have uncontrolled asthma that

  * might require bursts of oral or systemic corticosteroids, or
  * required the following due to ≥1 exacerbations within 12 months before baseline

    * systemic (oral and/or parenteral) corticosteroid treatment, or
    * hospitalization for >24 hours.
* Have known liver cirrhosis and/or chronic hepatitis of any etiology.
* Had Dupilumab treatment within 4 weeks prior to baseline
* Had prior treatment with tralokinumab.
* Treatment with topical agents: corticosteroids, calcineurin inhibitors, Janus Kinase (JAK) inhibitors, or phosphodiesterase-4 inhibitors, such as crisaborole within 2 weeks prior to baseline
* Treatment with any of the following agents within 4 weeks prior to the baseline

  * systemic immunosuppressive or immunomodulating drugs (e.g., systemic corticosteroids, cyclosporine, mycophenolate mofetil, IFN-gamma, azathioprine, methotrexate, and other immunosuppressants)
  * small molecules (e.g. JAK inhibitors)
  * phototherapy and photochemotherapy for AD

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2022-12-19 (Actual); Primary Completion 2024-01-11 (Actual); Study Completion 2025-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (37):
- United States (37):
  - River Region Dermatology and Laser, Montgomery, Alabama
  - Medical Dermatology Specialists, Phoenix, Arizona
  - First OC Dermatology, Fountain Valley, California
  - Axon Clinical Research, Inglewood, California
  - Avance Clinical Trials Inc, Laguna Niguel, California
  - Dermatology Research Associates, Los Angeles, California
  - Wallace Medical Group, Inc., Los Angeles, California
  - Clinical Science Institute, Santa Monica, California
  - Cura Clinical Research, Sherman Oaks, California
  - UConn Health, Farmington, Connecticut
  - Encore Medical Research of Boynton Beach, Boynton Beach, Florida
  - Total Vein and Skin LLC, Boynton Beach, Florida
  - Direct Helpers Research Center, Hialeah, Florida
  - Hollywood Dermatology, Hollywood, Florida
  - Miami Dermatology and Laser Research, Miami, Florida
  - Ziaderm Research, LLC., North Miami Beach, Florida
  - Olympian Clinical Research, Tampa, Florida
  - Skin Care Physicians of Georgia, Macon, Georgia
  - Advanced Medical Research, Sandy Springs, Georgia
  - Dundee Dermatology, West Dundee, Illinois
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Dermatology and Advanced Aesthetics, Lake Charles, Louisiana
  - Dermatology and Skin Cancer Specialists, LLC, Rockville, Maryland
  - Allcutis Research, Inc., Beverly, Massachusetts
  - Oakland Hills Dermatology, Auburn Hills, Michigan
  - The Derm Institute of West Michigan, Caledonia, Michigan
  - Revival Research Institute - Troy, Troy, Michigan
  - MediSearch Clinical Trials, Saint Joseph, Missouri
  - Allcutis Research, Inc, Portsmouth, New Hampshire
  - Windsor Dermatology, P.C., East Windsor, New Jersey
  - Sadick Research Group, New York, New York
  - OptiSkin Medical, New York, New York
  - Dermatologists of Greater Columbus, Bexley, Ohio
  - Dermatology and Skin Surgery Center, PC, Exton, Pennsylvania
  - Clinical Partners, LLC, Johnston, Rhode Island
  - Complete Dermatology, Sugar Land, Texas
  - Spokane Dermatology Clinic, Spokane, Washington

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- [Derived] Silverberg JI, Ackerman L, Bagel J, Stein Gold L, Blauvelt A, Rosmarin D, Chovatiya R, Zirwas M, Yosipovitch G, Waibel J, Murase JE, Lockshin B, Weisman J, Atwater AR, Proper J, Silk M, Pierce E, Piruzeli MLB, Montmayeur S, Schuster C, Zhong J, Rueda MJ, Pillai S, Simpson E. Lebrikizumab Improves Clinical Manifestations, Symptoms, and Quality of Life in Patients with Moderate-to-Severe Atopic Dermatitis Previously Treated with Dupilumab: Results from the ADapt Study. Dermatol Ther (Heidelb). 2026 Jan 19. doi: 10.1007/s13555-025-01644-3. Online ahead of print. PMID 41553700
- See also: A Study of Lebrikizumab (LY3650150) in Adult and Adolescent Participants With Moderate-to-Severe Atopic Dermatitis Previously Treated With Dupilumab — https://trials.lilly.com/en-US/trial/343315

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Results for maximum extended enrollment (ME2) participants will be posted after the study completion.
Groups:
- Lebrikizumab 250 mg Q2W: Participants received a 500 milligram (mg) loading dose of Lebrikizumab subcutaneously (SC) once every 2 weeks (Q2W) at baseline and Week 2, followed by 250 mg SC once Q2W until Week 16.
- Lebrikizumab 250 mg Q2W to Lebrikizumab 250 mg Q2W: Participants who received Lebrikizumab 250 mg SC once Q2W until Week 16 and who did not achieve IGA 0 or 1 (clear or almost clear) or a 75% reduction in the EASI score from baseline (EASI-75) at Week 16 continued to receive 250 mg SC once Q2W until Week 24.
- Lebrikizumab 250 mg Q2W to Lebrikizumab 250 mg Q4W: Participants who received Lebrikizumab 250 mg SC once Q2W until Week 16 and who achieved IGA 0 or 1 (clear or almost clear) or a 75% reduction in the EASI score from baseline (EASI-75) at Week 16, received 250 mg once every 4 weeks (Q4W) until Week 24.
Period: Treatment Period 1: Week 0 to Week 16
Arm/Group | Lebrikizumab 250 mg Q2W | Lebrikizumab 250 mg Q2W to Lebrikizumab 250 mg Q2W | Lebrikizumab 250 mg Q2W to Lebrikizumab 250 mg Q4W
Started | 86 | 0 | 0
Received at Least One Dose of Drug | 86 | 0 | 0
Intent-to-Treat (ITT) Population | 86 | 0 | 0
Completed | 59 | 0 | 0
Not Completed | 27 | 0 | 0
Not completed — Adverse Event | 5 | 0 | 0
Not completed — Protocol Deviation | 1 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Withdrawal by Subject | 12 | 0 | 0
Not completed — Physician Decision | 2 | 0 | 0
Not completed — Lost to Follow-up | 4 | 0 | 0
Not completed — Participant enrolled but didn't meet inclusion criteria 11 | 1 | 0 | 0
Not completed — Participant enrolled but did not meet inclusion criteria 3 | 1 | 0 | 0
Period: Treatment Period 2: Weeks 16 to Week 24
Arm/Group | Lebrikizumab 250 mg Q2W | Lebrikizumab 250 mg Q2W to Lebrikizumab 250 mg Q2W | Lebrikizumab 250 mg Q2W to Lebrikizumab 250 mg Q4W
Started (Treatment Period 2 Population: All enrolled patients who received at least 1 confirmed dose of 250 mg lebrikizumab during Weeks 16 to 24 of the Treatment Period.) | 0 | 18 | 41
Completed | 0 | 15 | 37
Not Completed | 0 | 3 | 4
Not completed — Protocol Deviation | 0 | 1 | 4
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population included all enrolled participants according to their planned intervention.
Groups:
- Lebrikizumab 250mg Q2W: Participants received a 500 mg loading dose of Lebrikizumab SC once Q2W at baseline and Week 2, followed by 250 mg SC once Q2W until Week 16. Responders who achieved IGA 0 or 1 (clear or almost clear) or a 75% reduction in the EASI score from baseline at Week 16 received 250 mg SC once Q4W until Week 24. Inadequate responders at Week 16 continued to receive 250 mg SC once Q2W until Week 24.
Arm/Group | Lebrikizumab 250mg Q2W
Number analyzed (Participants) | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.4 (20.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15
  Not Hispanic or Latino | 69
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 22
  White | 57
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 86

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Eczema Area and Severity Index 75 (EASI75) at Week 16
Description: The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent and clinical signs affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 to 72 (severe). The EASI75 responder is defined as a ≥ 75% improvement from baseline in the EASI score.
Time Frame: Week 16
Population: ITT population included all enrolled participants according to their planned intervention and had Week 16 EASI 75 data. Observed Cases (OC) analysis is applied here, where analysis is using all the observed data at each time point.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Lebrikizumab 250mg Q2W
Number analyzed (Participants) | 61
percentage of participants | 57.4 [46.9 to 67.3]

2. Secondary Outcome: Percentage of Participants Achieving EASI 75 at Week 24
Description: as for outcome 1
Time Frame: Week 24
Population: Population included all enrolled patients who received at least 1 confirmed dose of 250 mg lebrikizumab during Weeks 0 to 24 of the treatment period and had Week 24 EASI 75 data. OC analysis is applied here, where analysis is using all the observed data at each time point.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Lebrikizumab 250 mg Q2W to Lebrikizumab 250 mg Q2W: Participants who received Lebrikizumab 250 mg SC once Q2W until Week 16 and who did not achieve IGA 0 or 1 (clear or almost clear) or a 75% reduction in the EASI score from baseline (EASI-75) at Week 16, continued to receive 250 mg SC once Q2W until Week 24.
Arm/Group | Lebrikizumab 250 mg Q2W to Lebrikizumab 250 mg Q2W | Lebrikizumab 250 mg Q2W to Lebrikizumab 250 mg Q4W
Number analyzed (Participants) | 16 | 39
percentage of participants | 31.3 [16.1 to 51.8] | 71.8 [58.8 to 81.9]

3. Secondary Outcome: Percentage of Participants With an Investigator's Global Assessment (IGA) Score of 0 or 1 and a Reduction ≥2 Points From Baseline to Week 16
Description: The IGA measures the investigator's global assessment of the participant's overall severity of their AD, based on a static, numeric 5-point scale from 0 (clear skin) to 4 (severe disease). The score is based on the descriptors that best describe the overall appearance of the lesions at a given time point.
Time Frame: Baseline to Week 16
Population: ITT population included all enrolled participants according to their planned intervention and had Baseline IGA of at least 2. OC analysis is applied here, where analysis is using all the observed data at each time point.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Lebrikizumab 250mg Q2W
Number analyzed (Participants) | 62
percentage of participants | 38.7 [29.2 to 49.2]

4. Secondary Outcome: Percentage of Participants With an IGA Score of 0 or 1 and a Reduction ≥2 Points From Baseline to Week 24
Description: as for outcome 3
Time Frame: Baseline to Week 24
Population: Population included all enrolled patients who received at least 1 confirmed dose of 250 mg lebrikizumab during Weeks 0 to 24 of the treatment period and had Week 24 IGA score data. OC analysis is applied here, where analysis is using all the observed data at each time point.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Lebrikizumab 250 mg Q2W to Lebrikizumab 250 mg Q4W: Participants who received Lebrikizumab 250 mg SC once Q2W until Week 16 and who achieved IGA 0 or 1 (clear or almost clear) or a 75% reduction in the EASI score from baseline (EASI-75) at Week 16, received 250 mg Q4W until Week 24.
Arm/Group | Lebrikizumab 250 mg Q2W to Lebrikizumab 250 mg Q2W | Lebrikizumab 250 mg Q2W to Lebrikizumab 250 mg Q4W
Number analyzed (Participants) | 16 | 39
percentage of participants | 12.5 [4.2 to 31.6] | 48.7 [36.1 to 61.5]

5. Secondary Outcome: Percentage Change From Baseline in EASI Total Score From Baseline to Week 16
Description: The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent and clinical signs affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 to 72 (severe).
Time Frame: Baseline, Week 16
Population: ITT population included all enrolled participants according to their planned intervention and had Week 16 EASI data. OC analysis is applied here, where analysis is using all the observed data at each time point.
Measure: Mean (Standard Deviation); unit: percentage change
Groups:
- Lebrikizumab 250 mg Q2W: Participants received a 500 mg loading dose of Lebrikizumab SC once Q2W at baseline and Week 2, followed by 250 mg SC once Q2W until Week 16. Responders who achieved IGA 0 or 1 (clear or almost clear) or a 75% reduction in the EASI score from baseline at Week 16 received 250 mg SC once Q4W until Week 24. Inadequate responders at Week 16 continued to receive 250 mg SC once Q2W until Week 24.
Arm/Group | Lebrikizumab 250 mg Q2W
Number analyzed (Participants) | 61
percentage change | -73.3 (23.06)

6. Secondary Outcome: Percentage Change From Baseline in EASI Score From Baseline to Week 24
Description: as for outcome 5
Time Frame: Baseline, Week 24
Population: Population included all enrolled patients who received at least 1 confirmed dose of 250 mg lebrikizumab during Weeks 0 to 24 of the treatment period and had EASI score data. OC analysis is applied here, where analysis is using all the observed data at each time point.
Measure: Mean (Standard Deviation); unit: percentage change
Groups:
- Lebrikizumab 250 mg Q2W to Lebrikizumab 250 mg Q4W: Participants who received Lebrikizumab 250 mg SC once Q2W until Week 16 and who achieved IGA 0 or 1 (clear or almost clear) or a 75% reduction in the EASI score from baseline (EASI-75) at Week 16, received 250 mg once Q4W until Week 24.
Arm/Group | Lebrikizumab 250 mg Q2W to Lebrikizumab 250 mg Q2W | Lebrikizumab 250 mg Q2W to Lebrikizumab 250 mg Q4W
Number analyzed (Participants) | 16 | 39
percentage change | -64.6 (23.26) | -82.4 (15.93)

7. Secondary Outcome: Change From Baseline in EASI Score From Baseline to Week 16
Description: as for outcome 5
Time Frame: Baseline, Week 16
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lebrikizumab 250mg Q2W
Number analyzed (Participants) | 61
score on a scale | -17.4 (9.34)

8. Secondary Outcome: Change From Baseline in EASI Score From Baseline to Week 24
Description: as for outcome 5
Time Frame: Baseline, Week 24
Population: Population included all enrolled patients who received at least 1 confirmed dose of 250 mg lebrikizumab during Weeks 0 to 24 of the treatment period and had Week 24 EASI score data. OC analysis is applied here, where analysis is using all the observed data at each time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lebrikizumab 250 mg Q2W to Lebrikizumab 250 mg Q2W | Lebrikizumab 250 mg Q2W to Lebrikizumab 250 mg Q4W
Number analyzed (Participants) | 16 | 39
score on a scale | -17.4 (8.90) | -19.0 (8.29)

9. Secondary Outcome: Percentage of Participants Achieving EASI-90 (≥90% Reduction in EASI Score) From Baseline to Week 16
Description: The EASI assesses objective physician estimates of 2 dimensions of atopic dermatitis - disease extent and clinical signs affected: 0 = 0%; 1 = 1-9%; 2 = 10-29%; 3 = 30-49%; 4 = 50-69%; 5 = 70-89%; 6 = 90-100% and the severity of 4 clinical signs: (1) erythema, (2) edema/papulation, (3) excoriation, and (4) lichenification each on a scale of 0 to 3 (0 = none, absent; 1 = mild; 2 = moderate; 3 = severe) at 4 body sites (head/neck, trunk, upper limbs, and lower limbs). Half scores are allowed between severities 1, 2, and 3. The final EASI score was obtained by weight-averaging these 4 scores and will range from 0 to 72 (severe). The EASI90 responder is defined as a ≥ 90% improvement from baseline in the EASI score.
Time Frame: Baseline to Week 16
Population: ITT population included all enrolled participants according to their planned intervention and had Week 16 EASI 90 data. OC analysis is applied here, where analysis is using all the observed data at each time point.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Lebrikizumab 250mg Q2W
Number analyzed (Participants) | 61
percentage of participants | 29.5 [20.9 to 39.8]

10. Secondary Outcome: Percentage of Participants Achieving EASI-90 From Baseline to Week 24
Description: as for outcome 9
Time Frame: Baseline to Week 24
Population: Population included all enrolled patients who received at least 1 confirmed dose of 250 mg lebrikizumab during Weeks 0 to 24 of the treatment period and had Week 24 EASI 90 data. OC analysis is applied here, where analysis is using all the observed data at each time point.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Lebrikizumab 250 mg Q2W to Lebrikizumab 250 mg Q2W | Lebrikizumab 250 mg Q2W to Lebrikizumab 250 mg Q4W
Number analyzed (Participants) | 16 | 39
percentage of participants | 12.5 [4.2 to 31.6] | 35.9 [24.6 to 49.1]

11. Secondary Outcome: Percentage of Participants With a Pruritus Numeric Rating Scale (NRS) of ≥4 Points at Baseline Who Achieve at Least 4-point Reduction From Baseline to Week 16
Description: Pruritus NRS is an 11-point scale used by participants to rate their worst itch severity over the past 24 hours, with 0 indicating "No itch" and 10 indicating "Worst itch imaginable."
Time Frame: Baseline to Week 16
Population: ITT population included all enrolled participants according to their planned intervention and had a Baseline Pruritus NRS score of at least 4. OC analysis is applied here, where analysis is using all the observed data at each time point.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Lebrikizumab 250mg Q2W
Number analyzed (Participants) | 47
percentage of participants | 53.2 [41.4 to 64.7]

12. Secondary Outcome: Percentage of Participants With a Pruritus NRS of ≥4 Points at Baseline Who Achieve at Least 4-point Reduction From Baseline to Week 24
Description: as for outcome 11
Time Frame: Baseline to Week 24
Population: Population included all enrolled patients who received at least 1 confirmed dose of 250 mg lebrikizumab during Weeks 0 to 24 of the treatment period and had a >=4-point improvement from baseline in week 24 pruritus NRS score. OC analysis is applied here, where analysis is using all the observed data at each time point.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Lebrikizumab 250 mg Q2W to Lebrikizumab 250 mg Q2W | Lebrikizumab 250 mg Q2W to Lebrikizumab 250 mg Q4W
Number analyzed (Participants) | 13 | 26
percentage of participants | 53.8 [32.5 to 73.9] | 65.4 [49.3 to 78.6]

13. Secondary Outcome: Percentage of Participants With a Pruritus NRS of ≥3 Points at Baseline Who Achieve at Least 3-point Reduction From Baseline to Week 16
Description: as for outcome 11
Time Frame: Baseline to Week 16
Population: ITT population included all enrolled participants according to their planned intervention and had a Baseline Pruritus NRS score of at least 3. OC analysis is applied here, where analysis is using all the observed data at each time point.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Lebrikizumab 250mg Q2W
Number analyzed (Participants) | 48
percentage of participants | 72.9 [61.4 to 82.0]

14. Secondary Outcome: Percentage of Participants With a Pruritus NRS of ≥3 Points at Baseline Who Achieve at Least 3-point Reduction From Baseline to Week 24
Description: as for outcome 11
Time Frame: Baseline to Week 24
Population: Population included all enrolled patients who received at least 1 confirmed dose of 250 mg lebrikizumab during Weeks 0 to 24 of the treatment period and had a >=3-point improvement from baseline in week 24 pruritus NRS score. OC analysis is applied here, where analysis is using all the observed data at each time point.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Lebrikizumab 250 mg Q2W to Lebrikizumab 250 mg Q2W | Lebrikizumab 250 mg Q2W to Lebrikizumab 250 mg Q4W
Number analyzed (Participants) | 13 | 27
percentage of participants | 76.9 [54.2 to 90.4] | 77.8 [62.4 to 88.0]

15. Secondary Outcome: Percentage Change From Baseline in Pruritus NRS Score From Baseline to Week 16
Description: Pruritus NRS is an 11-point scale used by participants to rate their worst itch severity over the past 24 hours, with 0 indicating "No itch" and 10 indicating "Worst itch imaginable." Assessments were recorded daily by the participant using an electronic diary.
Time Frame: Baseline, Week 16
Population: ITT population included all enrolled participants according to their planned intervention and had week 16 pruritus NRS score. OC analysis is applied here, where analysis is using all the observed data at each time point.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Lebrikizumab 250mg Q2W
Number analyzed (Participants) | 53
percentage change | -55.6 (41.78)

16. Secondary Outcome: Percentage Change From Baseline in Pruritus NRS Score From Baseline to Week 24
Description: as for outcome 15
Time Frame: Baseline, Week 24
Population: Population included all enrolled patients who received at least 1 confirmed dose of 250 mg lebrikizumab during Weeks 0 to 24 of the treatment period and had week 24 pruritus NRS score. OC analysis is applied here, where analysis is using all the observed data at each time point.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Lebrikizumab 250 mg Q2W to Lebrikizumab 250 mg Q2W | Lebrikizumab 250 mg Q2W to Lebrikizumab 250 mg Q4W
Number analyzed (Participants) | 15 | 30
percentage change | -30.0 (99.07) | -62.0 (35.74)

17. Secondary Outcome: Percentage of Participants With a Sleep-Loss Scale of ≥2 Points at Baseline Who Achieve at Least 2-point Reduction From Baseline to Week 16
Description: Sleep loss due to interference of itch will be assessed by the participant. Participants rate their interference of itch on sleep based on a 5-point Likert scale [0 (not at all) to 4 (unable to sleep at all). Higher scores indicated a greater impact and worse outcome. Assessments will be recorded daily by the participant.
Time Frame: Baseline to Week 16
Population: ITT population included all enrolled participants according to their planned intervention and had a baseline Sleep-Loss scale score of at least 2. OC analysis is applied here, where analysis is using all the observed data at each time point.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Lebrikizumab 250mg Q2W
Number analyzed (Participants) | 24
percentage of participants | 41.7 [26.8 to 58.2]

18. Secondary Outcome: Percentage of Participants With a Sleep-Loss Scale of ≥2 Points at Baseline Who Achieve at Least 2-point Reduction From Baseline to Week 24
Description: as for outcome 17
Time Frame: Baseline to Week 24
Population: Population included all enrolled patients who received at least 1 confirmed dose of 250 mg lebrikizumab during Weeks 16 to 24 of the treatment period and had a >=2-point improvement from baseline in week 24 Sleep-Loss scale score. OC analysis is applied here, where analysis is using all the observed data at each time point.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Lebrikizumab 250 mg Q2W to Lebrikizumab 250 mg Q2W | Lebrikizumab 250 mg Q2W to Lebrikizumab 250 mg Q4W
Number analyzed (Participants) | 5 | 14
percentage of participants | 40.0 [14.3 to 72.8] | 42.9 [24.1 to 64.0]

19. Secondary Outcome: Change From Baseline in Sleep-Loss Scale From Baseline to Week 16
Description: as for outcome 17
Time Frame: Baseline, Week 16
Population: ITT population included all enrolled participants according to their planned intervention and had week 16 Sleep-Loss scale score. OC analysis is applied here, where analysis is using all the observed data at each time point.
Measure: Mean (Standard Deviation); unit: percentage of participants
Arm/Group | Lebrikizumab 250mg Q2W
Number analyzed (Participants) | 52
percentage of participants | -1.0 (1.00)

20. Secondary Outcome: Change From Baseline in Sleep-Loss Scale From Baseline to Week 24
Description: as for outcome 17
Time Frame: Baseline, Week 24
Population: Population included all enrolled patients who received at least 1 confirmed dose of 250 mg lebrikizumab during Weeks 0 to 24 of the treatment period and had week 24 Sleep-Loss scale score. OC analysis is applied here, where analysis is using all the observed data at each time point.
Measure: Mean (Standard Deviation); unit: percentage of participants
Arm/Group | Lebrikizumab 250 mg Q2W to Lebrikizumab 250 mg Q2W | Lebrikizumab 250 mg Q2W to Lebrikizumab 250 mg Q4W
Number analyzed (Participants) | 15 | 29
percentage of participants | -0.7 (1.07) | -1.1 (0.91)

21. Secondary Outcome: Change From Baseline in Skin Pain NRS From Baseline to Week 16
Description: The Skin Pain NRS is an 11-point scale used by participants to rate their worst level of skin pain over the past 24 hours, with 0 indicating "no pain" and 10 indicating "worst pain imaginable."
Time Frame: Baseline, Week 16
Population: ITT population included all enrolled participants according to their planned intervention and had week 16 skin pain NRS score. OC analysis is applied here, where analysis is using all the observed data at each time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lebrikizumab 250mg Q2W
Number analyzed (Participants) | 51
score on a scale | -3.2 (2.96)

22. Secondary Outcome: Change From Baseline in Skin Pain NRS From Baseline to Week 24
Description: as for outcome 21
Time Frame: Baseline, Week 24
Population: Population included all enrolled patients who received at least 1 confirmed dose of 250 mg lebrikizumab during Weeks 16 to 24 of the treatment period and had week 24 skin pain NRS score. OC analysis is applied here, where analysis is using all the observed data at each time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lebrikizumab 250 mg Q2W to Lebrikizumab 250 mg Q2W | Lebrikizumab 250 mg Q2W to Lebrikizumab 250 mg Q4W
Number analyzed (Participants) | 15 | 28
score on a scale | -2.8 (3.51) | -3.3 (2.73)

23. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) From Baseline to Week 16
Description: The DLQI questionnaire designed for participants aged >=16 years or more is a 10-item, validated questionnaire used to assess the impact of skin disease on the quality of life of an affected person. The 10 questions cover the following topics: symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment, over the previous week. Response categories include "Not at all," "A little," "A lot," and "Very much," with corresponding scores of 0, 1, 2, and 3 respectively. Questions 3-10 also have an additional response category of "Not relevant" which is scored as "0". Questions are scored from 0 to 3, giving a possible total score range from 0 (no impact of skin disease on quality of life) to 30 (maximum impact on quality of life). A high score is indicative of a poor quality of life.
Time Frame: Baseline, Week 16
Population: ITT population included all enrolled participants according to their planned intervention and had week 16 DLQI score. OC analysis is applied here, where analysis is using all the observed data at each time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lebrikizumab 250mg Q2W
Number analyzed (Participants) | 57
score on a scale | -8.7 (6.98)

24. Secondary Outcome: Change From Baseline in DLQI From Baseline to Week 24
Description: The DLQI questionnaire for participants aged 16 and above is a 10-item tool used to assess the impact of skin disease on quality of life. The 10 questions cover topics: symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment over the previous week. Response categories include "not at all," "a little," "a lot," and "very much," with corresponding scores of 0, 1, 2, and 3, respectively. Questions 3-10 have an additional response category of "not relevant," which is scored as "0." Questions are scored from 0 to 3. Total score ranges from 0 (no impact) to 30 (maximum impact), with higher scores indicating poorer quality of life.
Time Frame: Baseline, Week 24
Population: Population included all enrolled patients who received at least 1 confirmed dose of 250 mg lebrikizumab during Weeks 16 to 24 of the treatment period and had week 24 DLQI score. OC analysis is applied here, where analysis is using all the observed data at each time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lebrikizumab 250 mg Q2W to Lebrikizumab 250 mg Q2W | Lebrikizumab 250 mg Q2W to Lebrikizumab 250 mg Q4W
Number analyzed (Participants) | 15 | 35
score on a scale | -7.5 (7.13) | -9.5 (5.83)

25. Secondary Outcome: Change From Baseline in Children's Dermatology Life Quality Index (CDLQI) From Baseline to Week 16
Description: The CDLQI questionnaire designed for participants aged <16 years and It consists of 10 items that are grouped into 6 domains: symptoms & feelings, leisure, school or holidays, personal relationships, sleep, & treatment. The scoring of each question is: Very much =3; Quite a lot = 2; Only a little = 1; Not at all = 0. CDLQI total score is calculated by summing all 10 items responses and has a range of 0 to 30 (higher scores are indicative of greater impairment).
Time Frame: Baseline, Week 16
Population: ITT population included all enrolled participants according to their planned intervention and had week 16 CDLQI score. OC analysis is applied here, where analysis is using all the observed data at each time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lebrikizumab 250mg Q2W
Number analyzed (Participants) | 4
score on a scale | -3.0 (7.96)

26. Secondary Outcome: Change From Baseline in CDLQI From Baseline to Week 24
Description: as for outcome 25
Time Frame: Baseline, Week 24
Population: Population included all enrolled patients who received at least 1 confirmed dose of 250 mg lebrikizumab during Weeks 0 to 24 of the treatment period and had week 24 cDLQI score. OC analysis is applied here, where analysis is using all the observed data at each time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lebrikizumab 250 mg Q2W to Lebrikizumab 250 mg Q2W | Lebrikizumab 250 mg Q2W to Lebrikizumab 250 mg Q4W
Number analyzed (Participants) | 1 | 3
score on a scale | -1.0 (NA) — Only 1 participant included in the analysis, therefore standard deviation is not calculable. | -3.3 (9.45)

27. Secondary Outcome: Percentage Change From Baseline in SCORing Atopic Dermatitis (SCORAD) From Baseline to Week 16
Description: SCORAD is validated tool for assessing the extent and intensity of AD, it consists of 3 components: A=extent of AD as a percentage of each defined body area and reported as sum of all areas, with maximum score of 100%. B=severity of 6 specific symptoms of AD (redness, swelling, oozing/crusting, excoriation, skin thickening/lichenification, dryness) assessed using following scale: none=0, mild=1, moderate=2, or severe=3 for maximum of 18 total points. C=subjective assessment of itch and sleeplessness recorded by participant on visual analog scale (VAS), where 0=no itch/no sleeplessness and 10=worst imaginable itch/sleeplessness with maximum score of 20. SCORAD total score is calculated: A/5+7*B/2+ C to give total score range of 0 to 103, where 0=no disease to 103=severe disease.
Time Frame: Baseline, Week 16
Population: ITT population included all enrolled participants according to their planned intervention and had week 16 SCORAD score. OC analysis is applied here, where analysis is using all the observed data at each time point.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Lebrikizumab 250mg Q2W
Number analyzed (Participants) | 61
percentage change | -55.7 (22.46)

28. Secondary Outcome: Percentage Change From Baseline in SCORAD From Baseline to Week 24
Description: SCORAD is a validated tool for assessing the extent and intensity of AD. It consists of three components: A) the extent of AD as a percentage of each body area, with a maximum score of 100%; B) the severity of six specific symptoms (redness, swelling, oozing/crusting, excoriation, skin thickening/lichenification, dryness) rated from 0 (none) to 3 (severe) for a maximum of 18 points; and C) the subjective assessment of itch and sleeplessness on a visual analog scale (VAS) from 0 (no itch/sleeplessness) to 10 (worst imaginable itch/sleeplessness) with a maximum score of 20. The total SCORAD score is calculated as A/5 + 7*B/2 + C, ranging from 0 (no disease) to 103 (severe disease).
Time Frame: Baseline, Week 24
Population: Population included all enrolled patients who received at least 1 confirmed dose of 250 mg lebrikizumab during Weeks 16 to 24 of the treatment period and had week 24 SCORAD score. OC analysis is applied here, where analysis is using all the observed data at each time point.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | Lebrikizumab 250 mg Q2W to Lebrikizumab 250 mg Q2W | Lebrikizumab 250 mg Q2W to Lebrikizumab 250 mg Q4W
Number analyzed (Participants) | 16 | 38
percentage change | -47.4 (27.07) | -60.1 (23.51)

ADVERSE EVENTS:
Time Frame: Baseline Up To 24 Weeks AE data from the safety follow-up period and the continuous access period will be reported during the final results posting.
Description: All enrolled participants who received at least one confirmed dose of 250 mg lebrikizumab.
Groups:
- Lebrikizumab 250 mg Q2W: Participants received 500 milligram (mg) loading dose of Lebrikizumab subcutaneously (SC) once every 2 weeks (Q2W) at baseline and Week 2, followed by 250 mg SC once Q2W until Week 16.
- Lebrikizumab 250 mg Q2W to Q2W: Participants who received Lebrikizumab 250 mg SC once Q2W until Week 16 and who did not achieve IGA 0 or 1 (clear or almost clear) or a 75% reduction in the EASI score from baseline (EASI-75) at Week 16, continued to receive 250 mg SC once Q2W until Week 24.
- Lebrikizumab 250 mg Q2W to Q4W: Participants who received Lebrikizumab 250 mg SC once Q2W until Week 16 and who achieved IGA 0 or 1 (clear or almost clear) or a 75% reduction in the EASI score from baseline (EASI-75) at Week 16, received 250 mg once every 4 weeks (Q4W) until Week 24.
Arm/Group | Lebrikizumab 250 mg Q2W | Lebrikizumab 250 mg Q2W to Q2W | Lebrikizumab 250 mg Q2W to Q4W
All-Cause Mortality (participants affected / at risk) | 0/86 | 0/18 | 0/41
Serious Adverse Events (participants affected / at risk) | 1/86 | 0/18 | 1/41
Other Adverse Events (participants affected / at risk) | 38/86 | 6/18 | 6/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lebrikizumab 250 mg Q2W (N=86) | Lebrikizumab 250 mg Q2W to Q2W (N=18) | Lebrikizumab 250 mg Q2W to Q4W (N=41)
Cerebral vascular occlusion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Rash morbilliform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lebrikizumab 250 mg Q2W (N=86) | Lebrikizumab 250 mg Q2W to Q2W (N=18) | Lebrikizumab 250 mg Q2W to Q4W (N=41)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Swelling of eyelid (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Tooth impacted (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 3 (3) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral abdominal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (2) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2023-04-27): https://cdn.clinicaltrials.gov/large-docs/03/NCT05369403/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-23): https://cdn.clinicaltrials.gov/large-docs/03/NCT05369403/SAP_001.pdf